CLINICAL TRIAL: NCT06730724
Title: Is Ultrasound Measurement of Thenar Muscle Cross-Sectional Area Useful in the Evaluation of Carpal Tunnel Syndrome?: A Controlled Study
Brief Title: Thenar Muscle Ultrasound in CTS Evaluation
Status: Not yet recruiting | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principle Investigator, Beylikduzu State Hospital
Other Study IDs: BeylikduzuStateH12
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Carpal tunnel syndrome: Patients with carpal tunnel syndrome
  Interventions: Other: No intervention
- Control group: Healthy controls without carpal tunnel syndrome
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study will include 20 patients aged 18-75 years who have been diagnosed with carpal tunnel syndrome (CTS) based on electrophysiological examinations performed within the last three months, as well as 20 healthy volunteers without a CTS diagnosis. Sociodemographic data such as age, gender, height, weight, and BMI will be recorded. Pinch grip strength will be evaluated using a Jamar pinch meter, and hand grip strength will be assessed using a Jamar dynamometer. Ultrasound will be used to measure the cross-sectional area and thickness of the thenar muscles as well as the cross-sectional area of the median nerve. Additionally, previous electrophysiological examination results will be recorded for the CTS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years.
* Diagnosed with carpal tunnel syndrome based on electrophysiological examination within the last 3 months.
* Healthy volunteers without a diagnosis of carpal tunnel syndrome.
* Volunteered to participate in the study.

Exclusion Criteria:

* Refusal to participate in the study.
* History of surgery due to carpal tunnel syndrome.
* Presence of neuromuscular diseases.
* Presence of advanced osteoarthritis.
* Presence of psychiatric disorders.
* Presence of cognitive impairments that may hinder study participation.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Carpal tunnel syndrome and healthy controls
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Thenar Muscle Cross-Sectional Area (Ultrasound) | 0 day
  Measurement of the cross-sectional area of the thenar muscles using ultrasound to determine muscle atrophy or changes associated with carpal tunnel syndrome.

SECONDARY OUTCOMES:
Thenar Muscle Thickness (Ultrasound) | 0 day
  Assessment of the thickness of the thenar muscles using ultrasound to evaluate structural changes in patients with CTS.
Median Nerve Cross-Sectional Area (Ultrasound) | 0 day
  Measurement of the median nerve's cross-sectional area using ultrasound, a parameter commonly associated with CTS diagnosis and severity.
Pinch Grip Strength | 0 day
  Evaluated using the Jamar pinch meter, this outcome measures the functional strength of the thumb and index finger, which may be impaired in CTS.
Hand Grip Strength | 0 day
  Assessed with a Jamar dynamometer, this outcome measures overall hand strength and provides insights into functional limitations caused by CTS.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Şirin Ahısha, Principal Investigator — Beylikdüzü State Hospital
Locations (1):
- Beylikdüzü State Hospital, Istanbul, Beylikdüzü, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No